CLINICAL TRIAL: NCT01326442
Title: Phase 3 Study of Vitamin D and Omega-3 Supplementation to Reduce Risk of Metabolic Syndrome
Brief Title: Vitamin D and Omega-3 Inhibit Metabolic Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Kelly Anne Meckling, PhD, Professor, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011MeckVitD
Record Dates: First submitted 2011-03-29; First posted 2011-03-30 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Type 2 Diabetes Mellitus; Hypertension; Hyperlipidemia; Obesity
Keywords: weight loss; overweight; body composition; visceral obesity; insulin; glucose tolerance; cholesterol; hypertriglyceridemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Hyperlipidemias; Obesity; Weight Loss; Overweight; Obesity, Abdominal; Insulin Resistance; Hypertriglyceridemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- diet only (Experimental): low glycemic index diet, calorie restricted with exercise 3 times per week.
  Interventions: Other: low glycemic diet
- supplemented (Active Comparator): 2000 IU vitamin D3 plus 1.8 g EPA + DHA
  Interventions: Other: low glycemic diet; Dietary Supplement: vitamin D omega-3

INTERVENTIONS:
Other: low glycemic diet — a low glycemic diet, calorie restricted with exercise sessions 3 times per week
Dietary Supplement: vitamin D omega-3 — 2000 IU vitamin D3 plus 1.8 g EPA + DHA per day for 16 weeks.
  Arms: supplemented

SUMMARY:
The study will test the hypothesis that supplementing the diet of subjects with Metabolic Syndrome with 2000 IU vitamin D and 1.8 g omega-3 fatty acids (EPA + DHA) per day, will facilitate weight loss, improve body composition and reduce metabolic and biochemical risk factors associated with type II diabetes and cardiovascular disease. Adult men and women who meet the International Diabetes Federation criteria for Metabolic Syndrome will be enrolled and embark on a 16 week diet and exercise intervention using a low glycemic index diet with or without the supplementary vitamin D and omega-3. Subjects will be counseled weekly and blood collected at weeks 0 and 16.

ELIGIBILITY:
Inclusion Criteria:

* must have Metabolic Syndrome as defined by International Diabetes Federation
* must be able to swallow tablets and capsules
* must be 18 years of age or older
* must be physically capable of moderate intensity exercise

Exclusion Criteria:

* pregnant or lactating
* vegetarian

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
body weight | up to 16 weeks
  body weight will be measured to nearest 0.5 kg weekly

SECONDARY OUTCOMES:
Blood pressure | up to 16 weeks
  systolic and diastolic blood pressure will be measured in duplicate, weekly
Blood lipids | up to 16 weeks
  blood lipids will be measured at baseline and after study completion.
Glucose homeostasis | up to 16 weeks
  fasting blood glucose, insulin, HbA1c, CRP, cytokines and inflammatory markers will be measured at weeks 0 and 16 of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly A Meckling, PhD, Principal Investigator — University of Guelph
Locations (1):
- University of Guelph, Guelph, Ontario, Canada